### **Protocol Title**

# **Evaluation of novel molecular assays for the detection of influenza virus**

## **Principal Investigator**

Dr. Kelvin To MBBS, FRCPath, FHKCPath, FRCP (Edin), MD

> Date: 10<sup>th</sup> January 2019 Protocol number: FluA\_20190110

#### 1. PROTOCOL SYNOPSIS

| Protocol title | Evaluation of novel molecular assays for the detection of influenza virus |
|---|---|
| Hypothesis | Our novel molecular assays for the detection of influenza A virus will be non-inferior to current molecular assays published by the World Health Organization and the US Centers for Disease Control and Prevention |
| Primary objective | To evaluate the sensitivity and specificity of different molecular assays |
| Clinical specimens | Nasopharyngeal and saliva specimens previously tested for influenza A virus |
| Study design | We will randomly retrieve archived nasopharyngeal and saliva specimens that were previously tested for influenza A virus using commercially available assays in our laboratory, tested for influenza A virus at the Public Health Laboratory Service Branch in Hong Kong. These specimens will be tested for influenza A virus by 4 different RT-PCR assays as listed below: 1. Our new RT-PCR assay targeting PB2 gene 2. Our new RT-PCR assay targeting NS gene 3. M gene RT-PCR published by the World Health Organization 4. M gene RT-PCR published by the US CDC. |
| Primary outcome | Results of different RT-PCR assays |
| Secondary outcome | Cycle threshold (Ct) value of different RT-PCR assays |
| Data analysis | Sensitivity, specificity, positive predictive value and negative predictive value will be determined |

#### 2. BACKGROUND

Seasonal influenza virus causes an estimated 0.3-0.6 million deaths per year. Avian influenza virus H5N1, H7N9 and H5N6 has fatality rate of over 30% [1-3]. Swine influenza viruses from pigs have also infected humans [4].

Molecular assays are now used routinely in the detection of influenza viruses. The M gene is often used as the target for all influenza A viruses because the nucleotide sequence of this gene is relatively conserved among all the influenza A viruses. The World Health Organization and the US Centers for Disease Control and Prevention (CDC) have published protocols for molecular detection of influenza A virus M gene [5, 6].

However, recent studies have shown that mutations in the M gene have led to a reduced sensitivity of RT-PCR assay targeting this gene [7, 8]. Therefore, it is important to use

alternative conserved genes as the target of RT-PCR. In this study, our aim is to evaluate two new RT-PCR assays that are based on PB2 and NS gene segment.

#### 3. STUDY OBJECTIVES

1. To evaluate the sensitivity and specificity of different molecular assays

#### 4. STUDY DESIGN

#### 4.1. Overall study design

We will randomly retrieve archived nasopharyngeal and saliva specimens that were previously tested for influenza A virus using commercially available assays in our laboratory, tested for influenza A virus at the Public Health Laboratory Service Branch in Hong Kong. These specimens will be tested for influenza A virus by 4 different RT-PCR assays as listed below:

- 1. Our new RT-PCR assay targeting PB2 gene
- 2. Our new RT-PCR assay targeting NS gene
- 3. M gene RT-PCR published by the World Health Organization
- 4. M gene RT-PCR published by the US CDC.

Sensitivity and specificity will be determined as we described previously [9].

#### 4.2. Outcome measurements

#### 4.2.1. Primary outcome measure

1. Results of different RT-PCR assays

#### 4.2.2 Secondary outcome measure:

1. Cycle threshold (Ct) value of different RT-PCR assays

#### 4.3. Confidentiality of data

The specimens will be tested in an anonymous manner.

#### 4.4. Archive of data

The investigator will retain all study documentation pertaining to the conduct of the study at the study site for a period of at least 5 years.

#### 4.5. Ethical endorsement

The use of archived clinical specimen for microbiological testing has been approved by the Institutional Review Board (IRB) of the University of Hong Kong and Hospital Authority.

#### 5. SELECTION OF CLINICAL SPECIMENS FOR TESTING

#### 5.1. Inclusion criteria

- 1. Nasopharyngeal or saliva specimens of patients in Queen Mary Hospital of Hong Kong
- 2. Tested for influenza A virus using a commercially available assay or by the Public Health Laboratory Services Branch in Hong Kong

#### **5.2** Exclusion criteria

1. Insufficient specimen volume

#### 6. STUDY PROCEDURES

# 6.1 Nucleic acid extraction and real-time reverse transcription-polymerase chain reaction (RT-PCR) for influenza A virus

Saliva and nasopharyngeal specimens will be subjected to total nucleic acid (TNA) extraction by NucliSENS easyMAG (BioMerieux, Boxtel, Netherlands) as we described previously [10]. Briefly, 250  $\mu$ L of each specimen will be mixed with lysing buffer. After extraction, the nucleic acids will be recovered using 55  $\mu$ L of elution buffer.

Monoplex real-time RT-PCR assays for influenza A virus will be performed using QuantiNova Probe RT-PCR Kit (QIAGEN, Hilden, Germany). The reagent mixture (20  $\mu$ L) will contain 1x QuantiNova Probe RT-PCR Master Mix, 1x QN Probe RT-Mix, 0.8  $\mu$ M of each forward and reverse primer, 0.2  $\mu$ M of probe and 5  $\mu$ L of TNA as the template. The thermal cycling conditions will be 10 min at 45 °C for reverse transcription, 5 min at 95 °C for PCR initial activation, and 50 cycles of 5 s at 95 °C and 30 s at 55 °C. All reactions will be performed using the LightCycler 480 Real-Time PCR System (Roche, Basel, Switzerland). The primers and probes for the M gene RT-PCR have been published by the WHO and the US CDC [5, 6].

#### 7. STATISTICAL METHODS

#### 7.1 Sample size

We will perform all 4 RT-PCR assays on a total of 320 specimens, including

- 80 nasopharyngeal specimens which tested positive for influenza A by commercially-available molecular assays or by testing performed at the Public Health Laboratory Services Branch in Hong Kong
- 80 nasopharyngeal specimens which tested negative for influenza A by commercially-available molecular assays or by testing performed at the Public Health Laboratory Services Branch in Hong Kong

- 80 saliva specimens which tested positive for influenza A by commercially-available molecular assays
- 80 saliva specimens which tested negative for influenza A by commercially-available molecular assays

The sample size is based on feasibility of the study

#### 7.2 Analysis of the study

Sensitivity, specificity, positive predictive value and negative predictive value will be calculated for

- 1. All specimens
- 2. Nasopharyngeal specimens only
- 3. Saliva specimens only

#### 8. REFERENCES

- To KK, Chan JF, Chen H, Li L, Yuen KY. The emergence of influenza a h7n9 in human beings 16 years after influenza a h5n1: A tale of two cities. *Lancet Infect Dis.* 2013; **13**: 809-821.
- To KK, Tsang AK, Chan JF, Cheng VC, Chen H, Yuen KY. Emergence in china of human disease due to avian influenza a(h10n8)--cause for concern? *J Infect*. 2014; **68**: 205-215.
- To KK, Ng KH, Que TL, et al. Avian influenza a h5n1 virus: A continuous threat to humans. *Emerg Microbes Infect*. 2012; 1: e25.
- Freidl GS, Meijer A, de Bruin E, et al. Influenza at the animal-human interface: A review of the literature for virological evidence of human infection with swine or avian influenza viruses other than a(h5n1). *Euro Surveill*. 2014; **19**.
- World Health Organization. Who information for the molecular detection of influenza viruses. Available at <a href="http://www.Who.Int/influenza/gisrs\_laboratory/who\_information\_for\_the\_molecular\_detection\_of\_influenza\_viruses\_20171023\_final.Pdf">http://www.Who.Int/influenza/gisrs\_laboratory/who\_information\_for\_the\_molecular\_detection\_of\_influenza\_viruses\_20171023\_final.Pdf</a>. Accessed on august 15, 2018. 2017.
- 6 Selvaraju SB, Selvarangan R. Evaluation of three influenza a and b real-time reverse transcription-pcr assays and a new 2009 h1n1 assay for detection of influenza viruses. *J Clin Microbiol*. 2010; **48**: 3870-3875.
- Stellrecht KA. History of matrix genes mutations within per target regions among circulating influenza h3n2 clades over ten-plus-years. *J Clin Virol*. 2018; **107**: 11-18.
- Yang JR, Kuo CY, Huang HY, et al. Newly emerging mutations in the matrix genes of the human influenza a(h1n1)pdm09 and a(h3n2) viruses reduce the detection sensitivity of real-time reverse transcription-pcr. *J Clin Microbiol*. 2014; **52**: 76-82.
- To KK, Yip CC, Lai CY, et al. Saliva as a diagnostic specimen for testing respiratory virus by a point-of-care molecular assay: A diagnostic validity study. *Clin Microbiol Infect*. 2018.

To KK, Lu L, Yip CC, et al. Additional molecular testing of saliva specimens improves the detection of respiratory viruses. *Emerg Microbes Infect*. 2017; **6**: e49.